CLINICAL TRIAL: NCT01713439
Title: Phase 1 Study of Chemokine and Cytokine Gene Modified Allogeneic Neuroblastoma Cells for Treatment of Relapsed/Refractory Neuroblastoma Using a Retroviral Vector (CYCHEALL)
Brief Title: Allogeneic Neuroblastoma Cells for Relapsed/ Refractory Neuroblastoma, CYCHEALL
Acronym: CYCHEALL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other); St. Jude Children's Research Hospital (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Director/Professor Center for Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-6441 CYCHEALL; CYCHEALL (Other: Baylor College of Medicine)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Neuroblastoma
Keywords: Relapsed/Refractory Neuroblastoma; Retroviral vector injections; Allogeneic neuroblastoma cells; Lymphotactin; Interleukin-2 (IL-2)
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Injection of allogeneic neuroblastoma cells (Experimental): Retrovirally transduced allogeneic neuroblastoma cell lines secreting the human interleukin-2 and lymphotactin genes are frozen and, when needed, are thawed, mixed and irradiated. Relapsed or refractory patients are then treated with a course of four injections of their gene-modified tumor cells according to the following schedule: The first two injections will be given at week 1 and week 2. Patients will then have a two-week rest and the remaining two injections will be given at week 4 and week 5. A complete evaluation for evidence of toxicity and response will be performed at week 8 after a 3 week rest. At the 8 week evaluation, in the absence of progressive disease requiring therapy without excessive toxicity and if more transduced cells are available, the patient will have the option to receive four additional SC injections each separated by 1 month at the higher of the two dosage levels they originally received.
  Interventions: Biological: Injection of allogeneic neuroblastoma cells

INTERVENTIONS:
Biological: Injection of allogeneic neuroblastoma cells — Patients will receive a fixed dose of IL-2 gene modified tumor cells (10^7/kg, 10^8 max) already shown to be safe from a previous protocol, and an escalating dose of Lptn transduced tumor cells, beginning at 10^4/kg and rising to 10^7/kg (10^8 max). Patients will be assigned to an appropriate dose level for injection # 1. Injection #2 will contain 10 times more Lptn transduced cells than injection #1, until the max dose (10^8) has been reached in the first injection. The dose of injections 3 through 8 will be the same as the dose of injection #2. Initial injection volumes will be <1ml and should be injected in a single site. Only if these first patients show no undue local toxicity (including tumor cell growth) will multiple injection sites be used for subsequent high cell-dose studies.

SUMMARY:
The patient's have neuroblastoma that has come back, or not gone away. The cancer is harder to treat now. The investigators would like the patient's to be in this research study to determine the safety and dosage of special cells that may make the patient's own immune system fight the cancer. To do this the investigators will put two special genes into neuroblastoma cancer cells that have been grown in the lab. The genes put in make the cancer cells produce lymphotactin, a natural substance that attracts immune system cells to the cancer, and IL-2 a natural substance that may help the immune system kill cancer cells. Some of these cells will then be put into the patient's body. Studies of cancers in animals and in cancer cells that are grown in laboratories suggest that substances like lymphotactin and IL-2 do help the body kill cancer cells. A treatment similar to this has been used in twelve children previously and similar treatments are being used in adults with other cancers. This is a research study. The investigators do not know the best amount of special cells to use, so different children will get different numbers of cells.

The purpose of this study is to learn the side effects and safe "dosage" of these special cells. Participation in this study will last for 15 years.

DETAILED DESCRIPTION:
The investigators have grown neuroblastoma cells in the laboratory and put into them two specially produced mouse viruses (retroviruses) that carry the lymphotactin and the IL-2 gene. These lymphotactin and IL-2 genes are meant to help the immune system fight the cancer. The modified cancer cells will be injected under the patient's skin. There will be four shots. The second and subsequent shots will have ten times as many cells producing lymphotactin as the first. The patient will normally have these shots as an outpatient. Depending on response (if the patient's cancer has stayed the same or gotten smaller), the patient may be able to have four more of these shots.

Tests during and after treatment:

If the patient's blood has not been tested for HIV, the virus that causes AIDS, then the investigators will need to do this test. If this virus is present, this research treatment cannot be used.

Before the second shot, and then again about 2 weeks later, the investigators will remove some of the modified cells from the patient's body and study them. This will be done by a skin biopsy at the place where the cells were injected. These tests are to see whether the changes made in the laboratory are killing cancer cells.

To study how the immunity is working in the patient's body blood samples will be taken two to four days after each injection. This may be repeated 5-7 days after each injection if the patient's doctor thinks that it is necessary. After the patient stops receiving the injections, the blood draws will need to be repeated once a month for a year, and then once a year for fifteen years.

The patient will need to come to the clinic on the days the investigators take blood and will need to be seen at Texas Children's Cancer Center at weekly intervals for 6 weeks, then every other week for 6 weeks, and then monthly for a year. Then the patient will be seen in clinic or contacted by study personnel once a year for 15 years. Additional visits may be necessary.

To see if this research treatment is working, CAT scans, MRIs, or bone scans (these are different types of x-rays)will be done. Investigators will also take a bone marrow biopsy (bone marrow will be removed by use of a needle so that it can be looked at under the microscope). These tests will be done prior to treatment and repeated eight weeks later. In addition, if the patient receives the second set of four injections, these tests will be repeated at six months. If the neuroblastoma is not responding (if it has gotten larger), the investigators will offer the patient treatment with chemotherapy and/or radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients under 21 years of age at diagnosis with recurrent, advanced stage neuroblastoma shall be eligible for this protocol.
* Patients must have a life expectancy of at least 8 weeks.
* Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study, and have an absolute lymphocyte and neutrophil count of >500/mm3 each.
* Patients must not be currently receiving any investigational agents or have not received any tumor vaccines within the previous six months.
* Patients must have bilirubin <1.5 mg%.
* Patients must have creatinine <1.5 mg/dl.
* Patients must have ECOG performance status of 0-2 as below:

Grade Activity

* 0 Up and about, no restriction.
* 1 Ambulatory, no strenuous activity.
* 2 Ambulatory, capable of self-care appropriate for age.Up and about >50% of time, but unable to carry out any physical activities or attend school.
* 3 Limited self-care only. Up and about <50% of time.
* 4 Disabled, no self care. Bedridden or confined to chair.
* Patients must be willing to utilize one of the more effective birth control methods during the study and for six(6) months after the study is concluded. The male partner should use a condom.
* Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.

Exclusion Criteria:

* Patients must not be HIV-positive.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 1997-12 (Actual); Primary Completion 2001-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety of up to four subcutaneous (SC) injections of allogeneic neuroblastoma cells which have been genetically modified by measuring adverse events. | 8 weeks
  The patients will be given four injections as per the protocol schedule with the evaluation at Week 8 (month 2). This will constitute a course and the evaluation of the dose limiting toxicity will be done during this course. Any patient having grade 4 toxicity or having progressive disease during the course will be considered a failure.
To assess the safety of up to eight (total) injections in patients who have received the first four injections without unacceptable toxicity and have evidence of stable disease or better after receiving these injections by measuring adverse events. | 6 months
  The second course consists of administering another four injections as per the protocol schedule and evaluating at week 24 (6 months). The second course is conditional upon patients completing the first course with acceptable toxicity. This means that there will be at least 5 patients eligible to receive the second course.

SECONDARY OUTCOMES:
To determine whether MHC restricted or unrestricted antitumor immune responses are induced by SC injection of modified allogeneic neuroblasts and the cell doses required to produce these effects measured by punch biopsies. | 3 weeks
  For all the patients punch biopsies at the injection site will be done. From this a qualitative assessment of number of CD4 or CD8 or both types of cells will be made in order to understand the immune response.
Assess the antitumor effect by routine clinical response evaluation by imaging. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malcom Brenner, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas